CLINICAL TRIAL: NCT04300933
Title: Effects of Electroencephalogram-based Neurofeedback on Cognition in Adults With Subject Cognitive Decline
Brief Title: Neurofeedback Intervention for Preclinical Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: XuanwuH 2 (Other)
Collaborators: Beijing Institute of Technology (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HanYingsc3
Record Dates: First submitted 2020-03-06; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease; Subjective Cognitive Decline; Neurofeedback; Electroencephalogram
Keywords: Subjective cognitive decline; Intervention; Neurofeedback
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback therapy (Experimental): Fifty participants conduct neurofeedback daily for 5 days.
  Interventions: Behavioral: Electroencephalogram-based neurofeedback

INTERVENTIONS:
Behavioral: Electroencephalogram-based neurofeedback — In this project, SCD participants will receive electroencephalogram-based neurofeedback therapy, once a day, for 5 days. Then, the investigators will compare their memory changes between baseline and post-therapy visits.

SUMMARY:
Alzheimer's disease (AD) is the most common form of neurodegenerative disorders leading to dementia. Currently, there has been no effective pharmacologic therapy for this disease. Electroencephalogram-based neurofeedback is considered as a potentially treatment strategy. In this project, the investigators aim to investigate the effectiveness of neurofeedback therapy on cognition for individuals with subjective cognitive decline (SCD). Participants will receive electroencephalogram-based neurofeedback therapy once a day for successive five days. Then, the investigators will evaluate the changes of memory function between baseline and post-therapy visits.

DETAILED DESCRIPTION:
Currently, there has been no effective therapy for Alzheimer's disease (AD). Electroencephalogram-based neurofeedback is now considered as a potentially intervention and may positively affect cognitive function for patients with AD. However, there are few existing studies involving the role of neurofeedback on cognition for subjective cognitive decline (SCD).

Fifty participants with SCD will be recruited in this clinical trial. At baseline, neuropsychological tests are conducted. Participants will receive electroencephalogram-based neurofeedback therapy once a day for successive five days. After that, the investigators will evaluate the changes of memory measures, which is the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* 50-79 years old, right-handed and Mandarin-speaking subjects;
* self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event;
* normal age-adjusted, gender-adjusted and education-adjusted performance on standardised cognitive tests;
* concerns (worries) associated with memory complaint;
* failure to meet the criteria for MCI or dementia

Exclusion Criteria:

* a history of stroke;
* major depression (Hamilton Depression Rating Scale score > 24 points);
* other central nervous system diseases that may cause cognitive impairment, such as Parkinson's disease, tumors, encephalitis and epilepsy;
* cognitive impairment caused by traumatic brain injury;
* systemic diseases, such as thyroid dysfunction, syphilis and HIV;
* a history of psychosis or congenital mental growth retardation.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes of Auditory Verbal Learning Test (AVLT) score | Five days
  After intervention for five days, the investigators will compare baseline and post-therapy memory changes based on Auditory Verbal Learning Test (AVLT) scale, in order to investigate the therapeutic effectiveness of neurofeedback. The scale of AVLT focuses on the memory domain, especially AVLT-long delayed memory, with cut- off points as 5 (50-59 years old), 4 (60-69 years old), 3 (70-79 years old) and AVLT-recognition, with cut-off points as 20 (50-59 years old), 19 (60-69 years old), 18 (70-79 years old). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Han, PhD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Department of Neurolgy, Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The information of neuropsychological tests will be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: When summary data are published or starting 6 months after publication.
Access Criteria: The information of neuropsychological tests data will be shared.